CLINICAL TRIAL: NCT02854085
Title: Art Therapy and Music Reminiscence Activity in the Prevention of Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Rathi Mahendran, Senior Consultant Psychiatrist, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-16-095
Record Dates: First submitted 2016-07-07; First posted 2016-08-03 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Prevention of Cognitive Decline; Art Therapy; Music Reminiscence Activity; Elderly
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Art Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Art Therapy (Experimental): Art Therapy, 24 sessions
  Interventions: Behavioral: Art Therapy
- Music Reminiscence Activity (Experimental): Music Reminiscence Activity, 24 sessions
  Interventions: Behavioral: Music Reminiscence Activity
- Control (No Intervention): Participants will not participate in either of the interventions and will continue life as usual.

INTERVENTIONS:
Behavioral: Art Therapy — The Art Therapy will consist of creating art pieces, narrating thoughts and inner experiences in relation to the pieces produced (2 sessions a month) and guided visits to the art gallery (one session a month) and art museum (one session a month); there will be 12 sessions weekly for 12 weeks. For the next 6 months, sessions will be fortnightly and consist of creating an art piece once a month alternating with a visit to either the art museum or gallery, once a month; there will be 12 sessions in 6 months. Each session will last 45 minutes and will begin with 5 minutes of mindful relaxation to help participants focus on the task ahead.
  Other Names: AT
  Arms: Art Therapy
Behavioral: Music Reminiscence Activity — Music Reminiscence activity will be held weekly for 12 weeks and fortnightly for 6 months. Each session will last 45 minutes and will begin with 5 minutes of mindful relaxation to help participants focus on the task ahead. Session will entail listening and watching music videos and discussing activities, events and experiences related to the music; additional prompts such as photographs may be used to facilitate therapy.
  Other Names: MRA
  Arms: Music Reminiscence Activity

SUMMARY:
The objective of this study is to determine the impact of Art Therapy and Music Reminiscence Activity on cognition in community living elderly with Mild Cognitive Impairment (DSM V: Mild Neurocognitive Disorder) using a randomized control design.

Specifically, the structural cerebral changes that occur with the two interventions and the extent to which the therapies may reverse cognitive impairment and/or prevent further cognitive decline, will be determined.

The hypothesis is that participants in both active intervention arms will perform better on neuropsychological tests of cognition and will show positive changes on functional imaging studies compared to controls who will not receive any intervention. Participants in the interventions will also have positive changes in blood biomarkers, enhanced psychological well-being and reductions in anxiety and depressive symptoms compared to the control group. No a priori hypotheses were developed as to whether Art Therapy or Music Reminiscence Activity is more effective as the comparison is exploratory.

DETAILED DESCRIPTION:
Participants: 90 community-living elderly, with mild cognitive impairment.

Interventions: Participants will be randomized into 3 arms: Art Therapy, Music Reminiscence Activity or a Control arm. Sessions will be conducted weekly for 3 months and fortnightly for 6 months. Each intervention session will last for 40 minutes. The Control group will not receive any intervention and continue their life as usual.

Assessments: Demographic data will be collected at baseline. Neuropsychological tests of cognitive functioning will be done at baseline, 3 months and 9 months. Anxiety and depressive symptoms will be assessed at the 3 time-points. Blood sampling will occur at all time points (except control group, only at baseline and 9 months). Participants will also undergo a task-free brain fMRI scan at baseline and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Older person between 60 and 85 years of age, living in the community and fulfills the operational criteria/definition of MCI:

  1. At least one age-education adjusted neuropsychological test Z score <-1.5
  2. Do not meet DSM V criteria for a Major Neurocognitive Disorder
  3. Memory/Cognitive complaint preferably corroborated by a reliable informant
  4. Intact Activities of Daily Living
* Functions independently
* Does not have dementia
* Able to travel to the data collection site on their own and participate in the activity

Exclusion Criteria:

* Those who do not meet the above inclusion criteria (ie. do not have a MCI diagnosis)
* Those with Dementia/Major Neurocognitive Disorder or Normal Ageing
* Presence of a neurological condition e.g. epilepsy, Parkinson Disease, stroke
* Presence of a major psychiatric disorder e.g. Major Depression, Psychoses
* Terminal illness e.g. cancer
* Presence of significant visual and/or hearing impairment and Color Blindness
* Participants in another intervention study at the same time

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Neuropsychological Test: Change from baseline in Rey Auditory Verbal Learning Test scores at 3 months and 9 months | Measured at Baseline, 3 months and 9 months
  Measure: Number of items from a list of 15 items participant is able to recall immediately and 30 minutes later.
Neuropsychological Test: Change from baseline in Digit Span Task scores at 3 months and 9 months | Measured at Baseline, 3 months and 9 months
  Digit Span Task [(Digit Span Forward (DSF) and Digit Span Backward (DSB)]
  DSF Measure: 1 point for each correct sub-item response, Minimum: 0; Maximum 16 DSB Measure: 1 point for each correct sub-item response, Minimum: 0; Maximum 14
Neuropsychological Test: Change from baseline in Colour Trails Test scores at 3 months and 9 months | Measured at Baseline, 3 months and 9 months
  Colour Trails Test (CTT) 1 and 2
  Measure: Time to completion, in seconds for Trial 1 and Trial 2. Time Limit: 240s
Neuropsychological Test: Change from baseline in Block Design Test scores at 3 months and 9 months | Measured at Baseline, 3 months and 9 months
  Block Design (sub-test of the Wechsler Adult Intelligence Scale Tests)
  Measure: Respective sub-item test scores, based on time of completion and accuracy; Maximum score: 68
Change from baseline fMRI scan at 3 months | Measured at Baseline and 3 months
  Task-free Functional Magnetic Resonance Imaging (fMRI) will be employed to examine changes in functional connectivity.

SECONDARY OUTCOMES:
Change from baseline telomere lengths at 3 months and 9 months | Measured at Baseline, 3 months and 9 months
  Blood investigations to detect changes in telomere length

CONTACTS AND LOCATIONS:
Overall Officials: Rathi Mahendran, MBBS, Principal Investigator — National University of Singapore
Locations (1):
- Training and Research Academy, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kua EH, R Mahendran, L Feng, XF Tan, TP Ng. Preventive Psychiatry in Late Life: Studies on Depression and Dementia from the Singapore gerontology Research program. Taiwanese J Psychiatry 2013;27(4):267-275.
- [Background] Rawtaer I, Mahendran R, Yu J, Fam J, Feng L, Kua EH. Psychosocial interventions with art, music, Tai Chi and mindfulness for subsyndromal depression and anxiety in older adults: A naturalistic study in Singapore. Asia Pac Psychiatry. 2015 Sep;7(3):240-50. doi: 10.1111/appy.12201. Epub 2015 Jul 15. PMID 26178378
- [Background] Fam J, Yu Sun, Yu Chen, Tien HS, Feng L, EH Kua, R Mahendran. The Effects of Mindfulness Practice on mild cognitive impairment: a resting state functional connectivity study. Submission Pending.
- [Background] Sink KM, Espeland MA, Castro CM, Church T, Cohen R, Dodson JA, Guralnik J, Hendrie HC, Jennings J, Katula J, Lopez OL, McDermott MM, Pahor M, Reid KF, Rushing J, Verghese J, Rapp S, Williamson JD; LIFE Study Investigators. Effect of a 24-Month Physical Activity Intervention vs Health Education on Cognitive Outcomes in Sedentary Older Adults: The LIFE Randomized Trial. JAMA. 2015 Aug 25;314(8):781-90. doi: 10.1001/jama.2015.9617. PMID 26305648
- [Background] Chew EY, Clemons TE, Agron E, Launer LJ, Grodstein F, Bernstein PS; Age-Related Eye Disease Study 2 (AREDS2) Research Group. Effect of Omega-3 Fatty Acids, Lutein/Zeaxanthin, or Other Nutrient Supplementation on Cognitive Function: The AREDS2 Randomized Clinical Trial. JAMA. 2015 Aug 25;314(8):791-801. doi: 10.1001/jama.2015.9677. PMID 26305649
- [Background] Chancellor B, Duncan A, Chatterjee A. Art therapy for Alzheimer's disease and other dementias. J Alzheimers Dis. 2014;39(1):1-11. doi: 10.3233/JAD-131295. PMID 24121964
- [Background] Subramaniam M, Chong SA, Vaingankar JA, Abdin E, Chua BY, Chua HC, Eng GK, Heng D, Hia SB, Huang W, Jeyagurunathana A, Kua J, Lee SP, Mahendran R, Magadi H, Malladi S, McCrone P, Pang S, Picco L, Sagayadevan V, Sambasivam R, Seng KH, Seow E, Shafie S, Shahwan S, Tan LL, Yap M, Zhang Y, Ng LL, Prince M. Prevalence of Dementia in People Aged 60 Years and Above: Results from the WiSE Study. J Alzheimers Dis. 2015;45(4):1127-38. doi: 10.3233/JAD-142769. PMID 25672767
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Forsman AK, Nordmyr J, Wahlbeck K. Psychosocial interventions for the promotion of mental health and the prevention of depression among older adults. Health Promot Int. 2011 Dec;26 Suppl 1:i85-107. doi: 10.1093/heapro/dar074. PMID 22079938
- [Background] Koepsell TD, Monsell SE. Reversion from mild cognitive impairment to normal or near-normal cognition: risk factors and prognosis. Neurology. 2012 Oct 9;79(15):1591-8. doi: 10.1212/WNL.0b013e31826e26b7. Epub 2012 Sep 26. PMID 23019264
- [Background] Hilal S, Ikram MK, Saini M, Tan CS, Catindig JA, Dong YH, Lim LB, Ting EY, Koo EH, Cheung CY, Qiu A, Wong TY, Chen CL, Venketasubramanian N. Prevalence of cognitive impairment in Chinese: epidemiology of dementia in Singapore study. J Neurol Neurosurg Psychiatry. 2013 Jun;84(6):686-92. doi: 10.1136/jnnp-2012-304080. Epub 2013 Feb 5. PMID 23385846
- [Background] Paradise M, McCade D, Hickie IB, Diamond K, Lewis SJ, Naismith SL. Caregiver burden in mild cognitive impairment. Aging Ment Health. 2015 Jan;19(1):72-8. doi: 10.1080/13607863.2014.915922. Epub 2014 May 28. PMID 24866046
- [Background] Burnside I, Haight B. Reminiscence and life review: therapeutic interventions for older people. Nurse Pract. 1994 Apr;19(4):55-61. doi: 10.1097/00006205-199404000-00011. PMID 8035962
- [Derived] Mahendran R, Gandhi M, Moorakonda RB, Wong J, Kanchi MM, Fam J, Rawtaer I, Kumar AP, Feng L, Kua EH. Art therapy is associated with sustained improvement in cognitive function in the elderly with mild neurocognitive disorder: findings from a pilot randomized controlled trial for art therapy and music reminiscence activity versus usual care. Trials. 2018 Nov 9;19(1):615. doi: 10.1186/s13063-018-2988-6. PMID 30413216
- [Derived] Mahendran R, Rawtaer I, Fam J, Wong J, Kumar AP, Gandhi M, Jing KX, Feng L, Kua EH. Art therapy and music reminiscence activity in the prevention of cognitive decline: study protocol for a randomized controlled trial. Trials. 2017 Jul 12;18(1):324. doi: 10.1186/s13063-017-2080-7. PMID 28701205